CLINICAL TRIAL: NCT04408807
Title: Stress Induced by Screening for Retinopathy of Prematurity - Should Speculum and Indentation Rather be Avoided
Acronym: stressROP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Asimina Mataftsi, Associate Professor in Ophthalmology, Paediatric Ophthalmology and Strabismus, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 414/08-05-2019
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Sun Protection Factor; Surgical Instruments

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): ROPEE screening with speculum-free fundoscopy
  Interventions: Other: Speculum-free (SpF) fundoscopy
- Control Group (Active Comparator): ROPEE screening with speculum fundoscopy
  Interventions: Other: Speculum (Sp) fundoscopy

INTERVENTIONS:
Other: Speculum-free (SpF) fundoscopy — Indirect ophthalmoscopy without the use of eyelid speculum and scleral indentation
  Arms: Study Group
Other: Speculum (Sp) fundoscopy — Indirect ophthalmoscopy with the use of eyelid speculum and scleral indentation
  Arms: Control Group

SUMMARY:
The purpose is to assess the hypothesis that indirect ophthalmoscopy for retinopathy of prematurity eye examination (ROPEE) screening without the use of a lid speculum and scleral indentation (speculum-free, SpF) is less painful/stressful than funduscopy with speculum (Sp) and scleral indentation.

DETAILED DESCRIPTION:
A prospective randomized cross-over study was conducted for the comparison of the two techniques of funduscopy for ROPEE screening, i.e. with (Sp) or without (SpF) the use of a speculum and indentor. A random number table was used to allocate participants into either a) receiving Sp funduscopy on their first and SpF on their second screening examination a week later, or b) receiving SpF first and Sp a week later.

ELIGIBILITY:
Inclusion Criteria:

Preterm neonates undergoing screening for ROP, i.e.

* with GA < 32weeks and/or BW < 1501grams
* infants of greater BW and GA with increased comorbidity, e.g. sepsis, prolonged need for oxygen supplementation etc., as judged by the attending neonatologist

Exclusion Criteria:

1. Severe clinical condition with unstable vital signs to the extent that stress is not desired and the examination need to be postponed.
2. Diagnosis of traumatic apoptosis of the corneal epithelium / corneal ulcer.
3. Neonates under sedative/analgesic treatment.
4. Intraventricular hemorrhage (III,IV degree), moderate/severe neurological impairment, other conditions that could alter pain response.

Ages: 30 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Premature Infant Pain Profile-Revised score (PIPP) | a) before the intervention [the effect of mydriasis (PIPP1)] b) at the end of the intervention [the effect of funduscopy (PIPP2)] c) 10-20 minutes after the intervention [the overall effect of the examination, i.e. mydriasis and funduscopy (PIPP3)]

SECONDARY OUTCOMES:
Crying score of the Bernese pain scale | During the examination
Adverse events including arrythmia/bradycardia, apnoea, increased oxygen demands and feed intolerance | During the examination and during the 24 hours after the examination
Adequacy of judging the presence of treatment-requiring ROP | At the end of ROPEE screening
Duration of fundoscopy | During the examination

CONTACTS AND LOCATIONS:
Locations (1):
- "Papageorgiou" Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dhaliwal CA, Wright E, McIntosh N, Dhaliwal K, Fleck BW. Pain in neonates during screening for retinopathy of prematurity using binocular indirect ophthalmoscopy and wide-field digital retinal imaging: a randomised comparison. Arch Dis Child Fetal Neonatal Ed. 2010 Mar;95(2):F146-8. doi: 10.1136/adc.2009.168971. Epub 2009 Oct 8. PMID 19815939
- [Background] Mukherjee AN, Watts P, Al-Madfai H, Manoj B, Roberts D. Impact of retinopathy of prematurity screening examination on cardiorespiratory indices: a comparison of indirect ophthalmoscopy and retcam imaging. Ophthalmology. 2006 Sep;113(9):1547-52. doi: 10.1016/j.ophtha.2006.03.056. Epub 2006 Jul 7. PMID 16828505
- [Background] Mehta M, Adams GG, Bunce C, Xing W, Hill M. Pilot study of the systemic effects of three different screening methods used for retinopathy of prematurity. Early Hum Dev. 2005 Apr;81(4):355-60. doi: 10.1016/j.earlhumdev.2004.09.005. Epub 2004 Dec 8. PMID 15814220
- [Background] Dhillon B, Wright E, Fleck BW. Screening for retinopathy of prematurity: are a lid speculum and scleral indentation necessary? J Pediatr Ophthalmol Strabismus. 1993 Nov-Dec;30(6):377-81. doi: 10.3928/0191-3913-19931101-08. PMID 8120743
- [Result] Mataftsi A, Lithoxopoulou M, Seliniotaki AK, Talimtzi P, Oustoglou E, Diamanti E, Soubasi V, Ziakas N, Haidich AB. Avoiding use of lid speculum and indentation reduced infantile stress during retinopathy of prematurity examinations. Acta Ophthalmol. 2022 Feb;100(1):e128-e134. doi: 10.1111/aos.15085. Epub 2021 Dec 23. PMID 34939742